CLINICAL TRIAL: NCT04363983
Title: Interaction Between Host, Microenvironment and Immunity on Gastrointestinal Neoplasms: A Retro-prospective Cohort Study
Brief Title: Interaction Between Host, Microenvironment and Immunity on Gastrointestinal Neoplasms
Acronym: HoMING
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2019-A03330-57
Record Dates: First submitted 2020-04-20; First posted 2020-04-27 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: Gastrointestinal Neoplasms
Keywords: gastrointestinal cancer; micro-environment; immunity; host; microbiota
MeSH Terms: conditions — Gastrointestinal Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Located/resected colorectal cancer (Active Comparator)
  Interventions: Biological: Blood sampling; Procedure: Liver biopsy; Biological: Stool collect
- Advanced colorectal cancer (Active Comparator)
  Interventions: Biological: Blood sampling; Biological: Stool collect
- Located/resected pancreatic cancer (Active Comparator)
  Interventions: Biological: Blood sampling; Procedure: Liver biopsy; Biological: Stool collect
- Advanced pancreatic cancer (Active Comparator)
  Interventions: Biological: Blood sampling; Biological: Stool collect
- Located/resected biliary tract cancer (Active Comparator)
  Interventions: Biological: Blood sampling; Procedure: Liver biopsy; Biological: Stool collect
- Advanced biliary tract cancer (Active Comparator)
  Interventions: Biological: Blood sampling; Biological: Stool collect
- Located/resected gastroesophageal cancer (Active Comparator)
  Interventions: Biological: Blood sampling; Procedure: Liver biopsy; Biological: Stool collect
- Advanced gastroesophageal cancer (Active Comparator)
  Interventions: Biological: Blood sampling; Biological: Stool collect
- Located/resected neuroendocrine cancer (Active Comparator)
  Interventions: Biological: Blood sampling; Procedure: Liver biopsy; Biological: Stool collect
- Advanced neuroendocrine cancer (Active Comparator)
  Interventions: Biological: Blood sampling; Biological: Stool collect

INTERVENTIONS:
Biological: Blood sampling — Blood collection (50 ml) will be performed for all patients at baseline, at 1 month post-operative for resected patients (+ at the end of neoadjuvant treatment / before surgery if patient receives neoadjuvant treatment), and at 2-3 months after the beginning of the treatments in patients with metastases (+ at each progression).
  Following analysis should be performed with
  * serum for protein assays and characterization analysis of cytokines, new tumor markers and micro-RNA ...;
  * plasma for protein assays and characterization analysis of micro-RNA, VEC (the content of proteins, RNA, micro-RNA and DNA) and metabolomics;
  * PBMC for flow cytometry analysis, isolation macrophages;
  * whole blood for circulating tumor DNA (mutations by NGS, ddPCR,…; methylation) and circulating tumor cells.
Procedure: Liver biopsy — An intraoperative liver biopsy will be performed at free edge of liver with a triangular sample for local resected patients.
  This biopsy will be done with scissors, then patients will receive intraoperative hemostasis with mono- or bipolar coagulation. This procedure will be under laparoscopy or laparotomy without extending standard processing time.
  This biopsy seeks to allow the evaluate liver modifications testifying the preparing for premetastatic niche, which would allow to identify the patients with risk for hepatic relapsing; the same analysis on the tumors will be performed.
  Arms: Located/resected biliary tract cancer; Located/resected colorectal cancer; Located/resected gastroesophageal cancer; Located/resected neuroendocrine cancer; Located/resected pancreatic cancer
Biological: Stool collect — Stool collection will be performed for all patients at baseline, at 1 month post-operative for resected patients (+ at the end of neoadjuvant treatment / before surgery if patient receives neoadjuvant treatment), and at 2-3 months after the beginning of the treatments in patients with metastases (+ at each progression).
  Analysis will be performed for microbiota and metabolism analysis.

SUMMARY:
The primary objective: association study of characteristics of tumoral microenvironment and immunity of digestive cancers with patients' overall survival (OS).

DETAILED DESCRIPTION:
The study aims to explore relationship between the molecular subgroups (DNA and RNA analysis), tumor microenvironment, host (immunity system, premetastatic niche, microbiota, metabolism) and survival (prognostic value), response (predictive value) and tolerance (toxicities) to conventional treatments or immunotherapies in digestive cancers, in particular, in colorectal cancer and pancreaticobiliary cancer.

This is a prognostic monocentric study which includes 2 parts:

* one retrospective observational cohort for which 150 eligible patients (who have being diagnosed between 1998 to 2020) will be entered in the cohort per year during 22 years targeting 3300 patients and
* one prospective interventional cohort in which 3000 patients (diagnosis will be done between 2020-2030) will be enrolled during 10 years. 10 years of follow-up for all patients. This cohort is non comparative, non randomized, non control.

The enrollment will last 10 years in Digestive Surgery Department, Ambroise Paré Hospital, APHP.

There is any change in management of patients' care who will participate to the study, all of the treatment modalities (i.e. surgery, chemotherapy, radiotherapy, immunotherapy, intra-arterial treatments and supportive care) are possible and choice of treatment will be made by investigator physician, after multidisciplinary meeting validation, and according to referential and recommendations of practice in department.

Statistic analysis

The statistic analysis will be performed and reported according to the international guidelines STROBE for the observational studies.

ELIGIBILITY:
Inclusion Criteria:

* Carcinoma of colorectal, pancreatic, biliary tract or gastro-oesophageal, or neuroendocrine digestive tumors with cytologically or histologically proven, regardless of the stage;
* Diagnosis between 1998 and 2030;
* Be >/= 18 years;
* Have obtained signed informed consent (exemption for dead patients);
* Affiliated to the French social security - welfare system in France (CMU included).

Exclusion Criteria:

* Patient under tutoraship or curatorship;
* Foreign patient under AME schema, a medical help from the state in France;
* Pregnant or breastfeeding women (for prospective study);
* Any clinical, psychological or social reason which should influence patient compliance with protocol, according to investigator;
* Patient refusal.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6300 (Estimated)
Dates: Start 2021-01-13 (Actual); Primary Completion 2031-01 (Estimated); Study Completion 2031-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | monthly up to 3 months
  The OS is defined as timeframe between beginning of treatment (date of surgery or 1st cure of chemotherapy/immunotherapy) and death (regardless of reason).
Overall survival (OS) | yearly up to 10 years
  The OS is defined as timeframe between beginning of treatment (date of surgery or 1st cure of chemotherapy/immunotherapy) and death (regardless of reason).

SECONDARY OUTCOMES:
Survival without disease (SWD) | at month 1, 2 and 3, then yearly up to 10 years
  The SWD is defined as timeframe between date of surgical treatment and appearance of cancer relapse, 2nd cancer diagnosis or death (regardless reason).
Survival without progression (SWP) | at month 1, 2 and 3, then yearly up to 10 years
  The SWP is defined as timeframe between the beginning of treatment (date of 1st cure of chemotherapy/immunotherapy or date of 1st session of radiotherapy) and the 1st progression or death (regardless reason).
  The response of tumor will be evaluated according to the RECIST v1.1, Choi (intra-arterial treatments, antiangiogenic therapy) and/or iRECIST (immunotherapies) and/or imaging examinations depending on the given treatments.

CONTACTS AND LOCATIONS:
Overall Officials: Frédérique PESCHAUD, MD, PhD, Principal Investigator — Digestive Surgery Department, Ambroise Paré Hospital, APHP; Cindy NEUZILLET, MD, Study Director — Digestive Surgery Department, Ambroise Paré Hospital, APHP
Locations (1):
- Digestive Surgery Department, Ambroise Paré Hospital, APHP, Boulogne-Billancourt, France

IPD SHARING:
Plan to Share IPD: No